CLINICAL TRIAL: NCT03760224
Title: Effectiveness of WhatsApp Online Group Discussion for Smoking Relapse Prevention: a Pragmatic Randomized Controlled Trial
Brief Title: Effectiveness of WhatsApp Online Group Discussion for Smoking Relapse Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Relapse Prevention 2018
Record Dates: First submitted 2018-10-12; First posted 2018-11-30 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-03

CONDITIONS: Smoking Cessation
Keywords: Intervention; WhatsApp; Smoking Cessation; Relapse Prevention; Group Disscussion
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): WhatsApp group will receive at least 3 messages each week and allow real-time group discussion for the intervention period (8 weeks).
  Interventions: Other: WhatsApp group
- Control (Active Comparator): The control group will receive 3 mobile phone text messages each week in the 8 weeks after recruitment. This will be a one way message and no real-time discussion will be available.
  Interventions: Other: SMS group

INTERVENTIONS:
Other: WhatsApp group — WhatsApp group will allow real-time group discussion for 8 weeks
  Arms: Intervention
Other: SMS group — SMS group for 8 weeks
  Arms: Control

SUMMARY:
This study aims to examine the effectiveness and cost-effectiveness of WhatsApp group discussion for smoking relapse prevention. To assess the effect due to treatment modality through the WhatsApp social group, the frequency and topics of the posts in each social group will be analysed and in each participant. The primary hypothesis is whether quitters who participate in the WhatsApp group discussion will have a higher prevalence of validated tobacco abstinence at 12-month follow-up than those who do not. The second hypothesis is that greater participation in the social groups, indicated by number of posts received, posted and/or viewed, was associated with higher likelihood to quit at 12-month. The third hypothesis is that the WhatsApp intervention for a recent quitter is a more cost-effective option for tobacco abstinence and prolonged survival when compared to the control group.

DETAILED DESCRIPTION:
Study design:

This is a 2-arm open-labelled pragmatic randomized controlled trial, by comparing the 12-month tobacco abstinence between the recent quitters who will join WhatsApp group discussion (Intervention group) and those who will not (Control group). A 1:1 randomised allocation will be used. The intervention content for both trial arms in the proposed trial will be the same and based on the US practice guidelines for smoking cessation, therefore the intervention effects due to the treatment content will be the same in both groups. Only the intervention platform (WhatsApp vs text messaging service) and the communication mode (one-way vs interactive) will be different between the 2 groups. This trial will be a pragmatic effectiveness trial to examine the effect of our intervention delivered under a real-life setting. A less stringent eligibility criteria will be applied for the subjects, unobtrusive measurement on adherence, and include all subjects in the final analysis regardless of intervention compliance of each subject.

Subjects:

Patients who are receiving the smoking cessation service in the smoking cessation clinic of the Queen Elizabeth Hospital, Tung Wah Groups of Hospital, Shau Kei Wan Jockey Club Outpatient Clinic, Sai Ying Pun Jockey Club Outpatient Clinic and Pok Oi Chinese medicine clinic. Smoking Cessation Service will be invited to go through the screening process. These clinics are under Hospital Authority (n=3), or are non-governmental organizations that are funded by the government (n=7). Patients with the following inclusion criteria will be invited to participate in the RCT and will proceed to the recruitment procedure and intervention phase (Phase 2).

1. Daily tobacco user before service intake
2. Aged 18 years or above
3. Have enrolled or re-enrolled in the smoking cessation treatment for no more than 8 weeks
4. Not using tobacco products (including traditional cigarettes and heat-not-burn tobacco products) for 3 to 30 days
5. Able to communicate in Cantonese/Mandarin and read Chinese
6. Have a smart phone with local network connection The 4th criterion will be used because our proposed RCT will target the quitters who have recently quit, and exclude those who will have maintained a longer period of abstinence.

Exclusion criteria:

* Do not use WhatsApp as communication tool and show no interest to use WhatsApp
* Have unstable physical or psychological conditions as advised by doctors or counsellor in charge
* Have become pregnant in the past 2 months If the smoker meet all eligibility except the abstinence (the 4th criterion), he/she will be introduced about our RCT and asked to sign a consent form that allowing the HKU research staff to contact him again for another screening in (Phase 1).

Procedures:

Recruitment:

During a usual smoking cessation counseling session, the clinic counsellor or onsite trial recruitment staff (TRS) will briefly introduce the importance of relapse prevention and our phone-based relapse prevention intervention to the patient. If the patient agree to join, the TRS will then assess the eligibility section on the consent form. Patients who meet all the eligibility criteria will (i) be introduced about the RCT that they will be randomized to either the intervention or control group, and will participate in all follow-up assessments; (ii) be asked to sign the consent form; (iii) fill in a baseline questionnaire; and (iv) receive a leaflet, a self-help booklet and a souvenir. The consented participant will proceed to the intervention phase (Phase 2) and will be informed group allocation (WhatsApp social group (Intervention group) or text messaging service (control group)), where the option of platform will be determined by a randomization procedure.

If participants meet all eligibility criteria in the first screening except the tobacco abstinence for 3 to 30 days, the recruitment staff will invite them to set a quit day and complete the above recruitment procedures, but not to be randomized at that time. TRS will contact the participant 3 days after the quit date, and re-assess the eligibility of the RCT. Then, the participant will complete a baseline questionnaire, and receive a leaflet, a self-help booklet and a souvenir which are the same as those given to patient who meet all criteria. These participants will proceed to Phase 1.

If the patient do not meet other eligibility criteria in the first screening, the TRS will only provide a booklet (which are the same as those given to recruited patient) to the patient. He/she will be regarded as recruitment failure.

Phase 1 (Telephone follow-up) The participants in Phase 1 will be contacted by TRS to confirm the abstinence status. If the participant has not smoked for 3 days, the individual will be asked again if he/she agrees to receive the phone-based relapse prevention intervention. If agree, the TRS will briefly introduce again the RCT, and complete a brief questionnaire on the telephone. Afterwards, the participant will proceed to the intervention phase (Phase 2). If the participant disagrees, TRS will ask if he/she likes to participate in the study. If the participant does not wish to participate in the study, then the individual consent form will be destroyed and will not be contacted.

If the participant has not quit smoking, the TRS will ask the participant to set a quit date again and ask his/her consent to be re-contacted for another telephone screening after the quit date. Patients who do not want to be re-contacted will be regarded as recruitment failure. Otherwise, the TRS will contact the participant again after the quit date.

Interventions (Phase 2) When the TRS (that has gone through training to be a WhatsApp group moderator) collects about 7 to 14 participants (who have met all eligibility criteria) every one or two weeks from all clinics, he/she will set up the WhatsApp group with them. Each WhatsApp group (about 50 groups in total) will allow real-time group discussion for 8 weeks. The participants will receive each week at least 3 text messages or videos from a moderator, which will be based on the six approaches delineated in "Treatments for the Recent Quitter" of the US Clinical Practice Guidelines on Treating Tobacco Use and Dependence. Based on the Positive Psychology theories, a framework of four principles to enhance the online group moderation: (1) Using active listening skills to understand the thoughts and feelings behind individual's sharing; (2) Showing sincere, immediate, specific, and concrete appreciation and gratitude towards their sharing; (3) Mindful awareness of the group dynamics and giving strategic reactions; (4) Enhancement of self-efficacy, sense of control and satisfaction among the individual. All messages will address the five common problems leading to smoking relapse delineated in "Treatments for the Recent Quitter" of the US Clinical Practice Guidelines on Treating Tobacco Use and Dependence (26), including (1) lack of support for cessation; (2) negative mood or depression; (3) strong prolonged withdrawal symptoms; (4) weight gain; and (5) smoking lapses. If any participant shares their lapse or relapse experience in the group, the moderator will engage other individual to provide appreciation and support, or, if that individual agreed, actively refer him/her to existing cessation services.

To ensure quality assurance and intervention fidelity, all moderators will be provided training of smoking cessation knowledge, and moderating skills to motivate individual to share in WhatsApp. Moderators will also be trained on Positive Psychology by psychologist and counsellors from United Christian Hospital, United Centre of Emotional Health and Positive Living. This would allow moderators to learn a more positive approach to the language use within the group discussion and ways to express gratitude. The control group will only receive 3 mobile phone text messages each week in the 8 weeks after recruitment. These messages will be similar to those received by the intervention group. Our intervention will not interrupt the services that all individual will be receiving in the cessation clinics.

Several measures will be used to protect the privacy of personal data and internet safety of joining the WhatsApp groups. First, male and female individual in the WhatsApp group will be separated into different WhatsApp groups to avoid the possibility of misconduct or harassment. Second, participants will be reassured that all the WhatsApp posts can only be read by the individual and the moderator in the group as stated in the consent form. The TRS will only analyse all the data and WhatsApp posts anonymously. Third, moderator will encourage all the participants in the WhatsApp groups to share and post messages in the group, and avoid 1-to-1 individual communication via any channels within the study period. The moderator will also encourage the individual to report if anyone violate this regulation, and, if so, may give warnings to that individual. If the participant severely violate this regulation, this may result in termination of their participation. The moderator will also monitor the group conversation and report any events of misusing the contact information in the WhatsApp to the lead PI. This can reduce the chance of any misconduct, harassment, sharing and spread of harmful programs or virus, and unauthorized marketing using the contact information. Fourth, to avoid any internet virus or harmful links, the moderators will remind the group members not to open any suspicious links and files via WhatsApp. Lastly, individual can withdraw from the intervention study anytime over the study period. In the pilot RCT, about 83.4% of the eligible individual agreed to participate in the WhatsApp social groups after informed the above ethical issues.

After the recruitment, TRS will immediately send the contact details of the participant to our research staff for the randomization procedures.

Randomization:

TRS will send the Information of all the participant to the research staff, who are responsible to randomly allocate the group assignment. The principal investigator will generate a list of random numbers (for each recruitment site) and a list of group allocation, using the rand function of Excel. TRS will assign group allocation to each participant based on the list, followed by the intervention delivery.

Allocation concealment:

All TRS and participants will be concealed to the group allocation at recruitment. This randomization procedure will be done by the research staff in the research office.

Blinding:

The participant and group moderators cannot and will not be blinded to the intervention. Assessors of the follow-up outcomes and the research analysts will not be involved in the recruitment and intervention delivery, and will be blinded to the group allocation (single blindness).

Follow-up:

All individuals will be followed up via telephone by an allocation-blinded interviewer at 3-, 6- and 12-month after the random group allocation. Only the individual who report abstinence in the past 7 days during the 6- and 12- month follow-up will be invited to provide samples of exhaled breath and/or saliva for biochemical validation at their residence, workplace, or nearby, as preferred by the quitters. The Bedfont Smokerlyzer and iScreen OFD Cotinine Saliva Test Kit will be used for validations. The validation takes very short time (3 minutes ) and is easy.

Sample size determination:

Our pilot RCT showed that the OR of the CO validated quit rates between the intervention and control group was 2.04 (95%CI 0.74-5.65) (Intervention: 26.0%, Control: 15.0%). Because our proposed RCT will recruit quitters who have recently quit, PI have conservatively estimated that the OR will be 1.70 (23.0% vs 15.0%). To detect a significant difference of quit rate with 2-tailed z-test by GPower 3.1 between the two groups with a power of 90% (to reduce type II error) and 5% significant level (type I error), 1,008 participantswill be needed in total (504 individual per group).

Data analyses

Statistical analysis:

Using intention-to-treat analysis, participants who are lost to follow-up or drop out will be treated as smokers with no changes in daily cigarette consumption. The odds ratio, risk difference, and 95% confidence interval will be used to compare the primary and secondary outcomes between the two trial groups. Number needed to treat (NNT), which shows the number of treated participants needed to have one additional quitter at 12-month, will be computed by taking the reciprocal of the risk difference between the two trial groups. Assuming the missing outcomes are dependent on observed data (missing at random), an analysis using the multiple imputation (MI) procedure to impute the missing data will be conducted as sensitivity analysis. On the assumption that there will be no heterogeneity of intervention effect across clinics, the primary analysis will be conducted using logistic regression with and without adjustment for baseline characteristics. The assumption of homogeneity will first be checked by testing the clinic by intervention interaction with clinic as a fixed effect in the logistic model. If there is evidence of heterogeneity (i.e. p-value < 0.1), an analysis by generalized linear mixed (GLM) model with clinic as a random effect will be used to summarize the intervention effect on the primary outcome. Number of posts received and posted by each participant will be documented, and then included in the final GLM model to assess their association with the cessation outcome. All data analysis will be done using IBM SPSS version 25.0.

Text mining of the WhatsApp groups:

All discussion content will be archived and anonymized to remove identifying personal information. Due to a huge number of messages from the 50 WhatsApp groups, an automatic, computational text mining and visualization of the dataset will be used for the content analysis. First, utilizing a lexicon of keywords derived from our qualitative analysis of the pilot RCT, a heatmap visualization will be developed to illustrate the prevalence of the discussion topics. Second, topic modelling will be applied to investigate emerging themes in our WhatsApp dataset, using the Mallet implementation of the Latent Dirichlet Allocation topic modelling algorithm. Topic modelling algorithms take as input a text dataset (in this case, the WhatsApp dataset), and output a set of topics (and their associated keywords) in addition to estimates of the proportion of each topic.

Qualitative interview

To collect opinions towards the WhatsApp group intervention, purposive sampling will be used to select 20 individuals from the intervention group including both sexes, all age groups and all smoking status at 12-month, to participate in a qualitative face-to-face or telephone interview after the intervention. An interview guide with open-ended and iterative questions was used to probe for more experiences from the interviewees. Each interview will be conducted by the PI and a trained research assistant, and will last about 30 to 60 minutes.

The interview content was transcribed verbatim in Chinese for further analysis. The qualitative interview transcripts will be analysed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of social groups. Lead PI and two trained research assistants first used the open-coding method to identify relevant content in the transcripts; next, the lead PI will classified all labelled content into several independent themes showing distinct features of the social groups. The results were then discussed and consolidated in the panel meetings with the Co-I.

Cost-effectiveness analysis :

Cost-effectiveness analysis will be undertaken to indicate whether the intervention will be more cost-effective or even cost-saving option for a quitter over a time horizon of one year (within trial period) and lifetime. Within and lifetime cost-effectiveness analyses will be populated based on the healthcare provider perspective.

Model parameters input will be identified through within trial data and a review of local and overseas literature, where necessary. Within trial cost-effectiveness of WhatsApp intervention versus control group will be evaluated using total costs, the number of tobacco abstinence and total QALYs over the study period. EQ-5D-5L utility data at baseline and follow-ups from trial will estimate QALYs in two groups using area under the curve technique. Lifetime cost-effectiveness will be performed via Markov modelling that will simulate the annual health status progression of subjects in either intervention or control group. Both the successful and unsuccessful quitters after the trial will be subject to the annual transition probability from a status of no diseases to lung cancer, cardiovascular diseases, and other diseases, and then mortality. Former smokers may be relapsed after abstinence. Discounting will only be applied to total costs and QALY calculation under the lifetime horizon. Sensitivity analyses will be conducted where each parameter will be set at plausible lower and upper bounds based on 95% confidence interval of estimates in above data analysis.

The incremental cost-effectiveness ratio (ICER) in terms of cost per an additional tobacco abstinence gained, life-years gained, or QALYs gained for the intervention group in comparison to the control group will be reported. The WhatsApp intervention will be considered as cost-effective if its ICER will be less than 3 times per capita gross domestic product in Hong Kong recommended by WHO or the potential ICER threshold in Hong Kong. The cost-effectiveness model will be built using Microsoft Excel or Treeage Pro software.

ELIGIBILITY:
Inclusion Criteria:

* Daily tobacco user before service intake
* Aged 18 years or above
* Have enrolled or re-enrolled in the smoking cessation treatment for no more than 8 weeks
* Not using tobacco products (including traditional cigarettes and heat-not-burn tobacco products) for 3 to 30 days
* Able to communicate in Cantonese/Mandarin and read Chinese
* Have a smart phone with local network connection

Exclusion Criteria:

* Do not use WhatsApp as communication tool and show no interest to use WhatsApp
* Have unstable physical or psychological conditions as advised by doctors or counsellor in charge
* Have become pregnant in the past 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 928 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 years

REFERENCES:
- [Background] Mackay JM, Bettcher DW, Minhas R, Schotte K. Successes and new emerging challenges in tobacco control: addressing the vector. Tob Control. 2012 Mar;21(2):77-9. doi: 10.1136/tobaccocontrol-2012-050433. No abstract available. PMID 22345225
- [Background] Lam TH. Absolute risk of tobacco deaths: one in two smokers will be killed by smoking: comment on "Smoking and all-cause mortality in older people". Arch Intern Med. 2012 Jun 11;172(11):845-6. doi: 10.1001/archinternmed.2012.1927. No abstract available. PMID 22688993
- [Background] Segan CJ, Borland R, Greenwood KM. Can transtheoretical model measures predict relapse from the action stage of change among ex-smokers who quit after calling a quitline? Addict Behav. 2006 Mar;31(3):414-28. doi: 10.1016/j.addbeh.2005.05.023. Epub 2005 Jul 7. PMID 16005158
- [Background] Ockene JK, Emmons KM, Mermelstein RJ, Perkins KA, Bonollo DS, Voorhees CC, Hollis JF. Relapse and maintenance issues for smoking cessation. Health Psychol. 2000 Jan;19(1S):17-31. doi: 10.1037/0278-6133.19.suppl1.17. PMID 10709945
- [Background] Agboola S, McNeill A, Coleman T, Leonardi Bee J. A systematic review of the effectiveness of smoking relapse prevention interventions for abstinent smokers. Addiction. 2010 Aug;105(8):1362-80. doi: 10.1111/j.1360-0443.2010.02996.x. PMID 20653619
- [Background] Coley HL, Sadasivam RS, Williams JH, Volkman JE, Schoenberger YM, Kohler CL, Sobko H, Ray MN, Allison JJ, Ford DE, Gilbert GH, Houston TK; National Dental PBRN and QUITPRIMO Collaborative Group. Crowdsourced peer- versus expert-written smoking-cessation messages. Am J Prev Med. 2013 Nov;45(5):543-50. doi: 10.1016/j.amepre.2013.07.004. PMID 24139766
- [Background] Struik LL, Baskerville NB. The role of Facebook in Crush the Crave, a mobile- and social media-based smoking cessation intervention: qualitative framework analysis of posts. J Med Internet Res. 2014 Jul 11;16(7):e170. doi: 10.2196/jmir.3189. PMID 25016998
- [Background] Whittaker R, McRobbie H, Bullen C, Borland R, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2012 Nov 14;11:CD006611. doi: 10.1002/14651858.CD006611.pub3. PMID 23152238
- [Background] Selby P, van Mierlo T, Voci SC, Parent D, Cunningham JA. Online social and professional support for smokers trying to quit: an exploration of first time posts from 2562 members. J Med Internet Res. 2010 Aug 18;12(3):e34. doi: 10.2196/jmir.1340. PMID 20719739
- [Background] Duke JC, Hansen H, Kim AE, Curry L, Allen J. The use of social media by state tobacco control programs to promote smoking cessation: a cross-sectional study. J Med Internet Res. 2014 Jul 10;16(7):e169. doi: 10.2196/jmir.3430. PMID 25014311
- [Background] Pechmann C, Delucchi K, Lakon CM, Prochaska JJ. Randomised controlled trial evaluation of Tweet2Quit: a social network quit-smoking intervention. Tob Control. 2017 Mar;26(2):188-194. doi: 10.1136/tobaccocontrol-2015-052768. Epub 2016 Feb 29. PMID 26928205
- [Background] Cheung YT, Chan CH, Lai CK, Chan WF, Wang MP, Li HC, Chan SS, Lam TH. Using WhatsApp and Facebook Online Social Groups for Smoking Relapse Prevention for Recent Quitters: A Pilot Pragmatic Cluster Randomized Controlled Trial. J Med Internet Res. 2015 Oct 22;17(10):e238. doi: 10.2196/jmir.4829. PMID 26494159
- [Background] Cheung YTD, Chan CHH, Wang MP, Li HCW, Lam TH. Online Social Support for the Prevention of Smoking Relapse: A Content Analysis of the WhatsApp and Facebook Social Groups. Telemed J E Health. 2017 Jun;23(6):507-516. doi: 10.1089/tmj.2016.0176. Epub 2016 Dec 2. PMID 27911654
- [Background] Hughes JR, Keely J, Naud S. Shape of the relapse curve and long-term abstinence among untreated smokers. Addiction. 2004 Jan;99(1):29-38. doi: 10.1111/j.1360-0443.2004.00540.x. PMID 14678060
- [Background] Chen AT, Zhu SH, Conway M. What Online Communities Can Tell Us About Electronic Cigarettes and Hookah Use: A Study Using Text Mining and Visualization Techniques. J Med Internet Res. 2015 Sep 29;17(9):e220. doi: 10.2196/jmir.4517. PMID 26420469
- [Background] Census & Statistics Department (Hong Kong SAR government). Thematic Household Survey, Report No. 59: Pattern of Smoking. Hong Kong: Census & Statistics Department 2016.
- [Background] World Health Organization. Parties to the WHO framework convention on tobacco control, 2012. http://www.who.int/fctc/signatories_parties/en/index.html#. Geneva: World Health Organization, 2012.
- [Background] Marlatt G, Gordon J. Determinants of relapse: implications for the maintenance of behavior change. In: Davidson PO, Davidson SM, editors. Behavioral Medicine: Changing Health Lifestyles. New York: Brunner/Mazel; 1980. p. 410 - 52.
- [Background] Phua J. Participating in Health Issue-Specific Social Networking Sites to Quit Smoking: How Does Online Social Interconnectedness Influence Smoking Cessation Self-Efficacy? J Commun. 2013;63(5):933-52. doi: 10.1111/jcom.12054.
- [Background] Fiore MC, Jaén CR, Baker TB, Bailey WC, Benowitz NL, Curry SJ, et al. Treating tobacco use and dependence: 2008 update. Rockvill: MD: Department of Health and Human Services, 2008.
- [Background] Snyder CR, Lopez SJ. Positive psychology : the scientific and practical explorations of human strengths Thousands Oaks, Calif: SAGE Publications; 2007.
- [Background] Blei DM, Ng AY, Jordan MI. Latent dirichlet allocation. J Mach Learn Res. 2003;3:993-1022.
- [Background] Blei DM. Probabilistic topic models. Commun ACM. 2012;55(4):77-84. doi: 10.1145/2133806.2133826.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on our pilot study, we calculated our sample size to be 1008 participants. As we predicted that there would be participants who fail to be contacted or fail to quit for 3 days, we recruited more than the target number of participants before the start of the intervention. Yet, due to the COVID-19, we recruited 928 participants and enrolled in the study.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 469 | 459
Completed | 469 | 459
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 469 | 459 | 928
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 443 | 434 | 877
  >=65 years | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.00 (11.70) | 42.97 (11.72) | 42.99 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 103 | 188
  Male | 384 | 356 | 740
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 469 | 459 | 928
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 469 | 459 | 928
Fagerstrom Test For Nicotine Dependence [Mean (Standard Deviation); unit: scores on a scale] — The total score ranged from 0 to 10. A higher score indicates the participants' more intense physical dependence on nicotine.
  scores on a scale | 5.1 (2.5) | 5.1 (2.6) | 5.1 (2.5)
Minnesota Nicotine Withdrawal Scale [Mean (Standard Deviation); unit: scores on a scale] — The total score ranged from 0 to 36. A higher score indicates participants had more withdrawal symptoms.
  scores on a scale | 18.1 (6.8) | 18.0 (7.0) | 18.1 (6.9)
Importance of quitting [Mean (Standard Deviation); unit: scores on a scale] — The importance of quitting will be evaluated on a scale of 0 to 10 (0, least important; 10, most important). For the scale of measuring quitting importance, higher scores mean a better outcome.
  scores on a scale | 8.4 (1.8) | 8.4 (1.6) | 8.4 (1.7)
Difficulty of quitting [Mean (Standard Deviation); unit: scores on a scale] — The difficulty of quitting will be evaluated on a scale of 0 to 10 (0, least difficult; 10, most difficult). For the scale of measuring quitting difficulty, higher scores mean a worse outcome.
  scores on a scale | 7.4 (2.2) | 7.4 (2.1) | 7.4 (2.2)
Confidence of quitting [Mean (Standard Deviation); unit: scores on a scale] — Confidence in quitting will be evaluated on a scale of 0 to 10 (0, least confident; 10, most confident). For the scale of measuring quitting confidence, higher scores mean a better outcome.
  scores on a scale | 6.4 (2.2) | 6.6 (2.2) | 6.5 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Passed the Biochemical Validated Abstinence at 12-month Follow-up
Description: Exhaled carbon monoxide below 4ppm using a Smokerlyzer, and a saliva cotinine 10ng/ml or below using the iScreen OFD Cotinine Saliva Test Kit
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 56 | 54

2. Secondary Outcome: Number of Participants Who Passed the Biochemical Validated Abstinence at 6-month Follow-up
Description: as for outcome 1
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 69 | 75

3. Secondary Outcome: Number of Participants Who Self-reported 7-day Abstinence at 3-month Follow-up
Description: Self-reported abstinence in the past 7 days at 3-month follow-up
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 256 | 257

4. Secondary Outcome: Number of Participants Self-reported 7-day Abstinence at 6-month Follow-up
Description: Self-reported abstinence in the past 7 days at 6-month follow-up
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 229 | 232

5. Secondary Outcome: Number of Participants Self-reported 7-day Abstinence at 12-month Follow-up
Description: Self-reported abstinence in the past 7 days at 12-month follow-up
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 200 | 216

6. Secondary Outcome: Number of Participants Who Reported Smoking Relapse at 3-month Follow-up
Description: Consuming 5 cigarettes or more in 3 consecutive days in the past 3 months
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 213 | 202

7. Secondary Outcome: Number of Participants Who Reported Smoking Relapse at 6-month Follow-up
Description: Consuming 5 cigarettes or more in 3 consecutive days in the past 6 months
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 240 | 227

8. Secondary Outcome: Number of Participants Who Reported Smoking Relapse at 12-month Follow-up
Description: Consuming 5 cigarettes or more in 3 consecutive days in the past 12 months
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 269 | 243

9. Secondary Outcome: Number of Participants Who Reported Self-reported Continuous Abstinence
Description: Self-reported continuous abstinence
Time Frame: 3 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 256 | 257

10. Secondary Outcome: Number of Participants Who Self-reported Continuous Abstinence
Description: Self-reported continuous abstinence
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 185 | 187

11. Secondary Outcome: Number of Participants Who Self-reported Continuous Abstinence
Description: Self-reported continuous abstinence
Time Frame: 12 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
Participants | 130 | 141

12. Other Pre Specified Outcome: Frequency of Smoking Urge
Description: Frequency (in the past week) of smoking urge will be evaluated according to their frequency of their smoking urges on a scale of 0 (none at all) to 4 (ever hour or more).
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 2.09 (1.21) | 2.13 (1.19)

13. Other Pre Specified Outcome: Intensity of Smoking Urge
Description: Intensity (in the past day) of smoking urge will be evaluated according to their intensity of their smoking urges on a scale of 1 (never have smoking urges) to 5 (smoking urges every hour or more).
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 1.70 (0.95) | 1.79 (1.02)

14. Other Pre Specified Outcome: Frequency of Smoking Urge
Description: as for outcome 12
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 1.72 (1.12) | 1.73 (1.05)

15. Other Pre Specified Outcome: Intensity of Smoking Urge
Description: as for outcome 13
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 1.46 (0.83) | 1.46 (0.78)

16. Other Pre Specified Outcome: Frequency of Smoking Urge
Description: as for outcome 12
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 2.04 (1.37) | 2.07 (1.46)

17. Other Pre Specified Outcome: Intensity of Smoking Urge
Description: as for outcome 13
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 1.37 (0.82) | 1.39 (0.83)

18. Other Pre Specified Outcome: EuroQoL 5-Dimension 5-Level (EQ-5D-5L)
Description: EuroQol 5-dimension 5 level (EQ-5D-5L) health utility scores on a 1 (No problem) -5 (unable or extreme pain/ anxious) scales which assess participants mobility, self care, usual activities, pain/ discomfort and their anxiety/ depression. After obtaining the data, results were re-calculated and transferred based on Hong Kong population norm. After calculation, the total score ranged from -0.864 to 1. Higher score indicates better health status. Calculations of this scale were based on Hong Kong population provided by Wong EL and colleagues (Wong EL, Ramos-Goni JM, Cheung AW, Wong AY, Rivero-Arias O. Assessing the use of a feedback module to model EQ-5D-5L health states values in Hong Kong. The Patient-Patient-Centered Outcomes Research. 2018 Apr;11(2):235-47.).
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 0.96 (0.13) | 0.97 (0.08)

19. Other Pre Specified Outcome: EuroQoL 5-Dimension 5-Level (EQ-5D-5L)
Description: as for outcome 18
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 0.96 (0.11) | 0.95 (0.11)

20. Other Pre Specified Outcome: EuroQoL 5-Dimension 5-Level (EQ-5D-5L)
Description: as for outcome 18
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 0.97 (0.09) | 0.97 (0.10)

21. Other Pre Specified Outcome: Change in Quality of Life Inventory
Description: Quality of Life Inventory (QoLI) , 7 items with 3-point rating scale for importance (1 not important, 3 very important), and 3-point rating scale for satisfaction (1 not satisfied, 3 very satisfied) in terms of health, economy, work, hobbies, relationship with partner, friendship and relationship with family.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
score on a scale | 2.45 (1.25) | 2.31 (1.36)

22. Other Pre Specified Outcome: Change in Quality of Life Inventory
Description: as for outcome 21
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
scores on a scale | 2.50 (1.30) | 2.46 (1.35)

23. Other Pre Specified Outcome: Nicotine Withdrawals
Description: Minnesota Nicotine Withdrawal Scale (MNWS) using Likert-type scale for the severity ratings, ranging from 0 (not at all) to 4 (severe) in terms of their desire and craving to smoke, insomnia, awakening at night, difficulty in concentration, anxious,depressed, restless and irritable. As the 9 items were rated from 0-4, therefore, the total score ranged from 0-36. A higher score indicates participants had more withdrawal symptoms.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
scores on a scale | 11.85 (3.88) | 12.37 (4.96)

24. Other Pre Specified Outcome: Nicotine Withdrawals
Description: as for outcome 23
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
scores on a scale | 11.30 (3.27) | 11.71 (4.14)

25. Other Pre Specified Outcome: Nicotine Withdrawals
Description: as for outcome 23
Time Frame: 12 month
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 469 | 459
scores on a scale | 10.90 (3.72) | 11.46 (4.24)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/469 | 0/459
Serious Adverse Events (participants affected / at risk) | 0/469 | 0/459
Other Adverse Events (participants affected / at risk) | 0/469 | 0/459

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03760224/Prot_SAP_001.pdf